CLINICAL TRIAL: NCT03129581
Title: Using Novel Digital Mobile Technology to Implement Time-restricted Feeding to Improve the Metabolic Health of Overweight and Obese Participants at Risk for Developing Diabetes
Brief Title: Metabolic Impact of Time Restricted Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2016-25155
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Diet Modification
Keywords: obesity, diet, sleep activity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: randomized, non-blinded, behavioral intervention pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted (Active Comparator): This group will receive dietary counseling.
  Interventions: Behavioral: Dietary Counseling
- Time Unrestricted (No Intervention): This group will not receive dietary counseling.

INTERVENTIONS:
Behavioral: Dietary Counseling — Counseling to only eat during a restricted amount of time.
  Arms: Time Restricted

SUMMARY:
The investigators are interested in how time-restricted feeding will impact weight, sleep duration and efficacy, and activity levels in obese adults. Significant advances in digital mobile technology allow detailed measures of an individual's habits, permitting the opportunity for personalized dietary and lifestyle recommendations. This is especially relevant as time-restricted feeding appears to promote weight loss independent of calorie intake, potentially shifting the paradigm of dietary recommendations from a calorie-based to a time-based perspective.

DETAILED DESCRIPTION:
Given the obesity epidemic, there is intense medical and public interest in dietary and lifestyle management to mitigate obesity and its associated complications. Although weight loss has traditionally focused on restricting calories, it is well described that most people are unable to maintain the caloric restriction required to long term weight loss or maintenance. This proposal will address whether restricting the timing of food intake, rather than restricting calories, may facilitate weight loss and provide metabolic benefits. It has been recently shown that the average American eats over the course of 15 hours per day. Such an eating cycle dictates that most people are always in a fed metabolic state and likely misaligns circadian patterns. Time-restricted feeding (TRF) is the process of limiting food consumption to a specific window of time (e.g. 8 hours per day) and is associated with weight loss in humans and metabolic improvements in rodent studies. Significant advances in digital mobile technology now allow further detailed measures of an individual's habits to facilitate this analysis. Thus, the objective of this study is to test the health related effects of 12 week TRF (8 hour fed and 16 hour fasting cycle) in overweight/obese adults. The investigators hypothesize that TRF will 1) improve sleep duration, sleep efficacy, increase activity and increase basal metabolic rate, 2) promote weight loss and lower body fat, and 3) improve insulin sensitivity and postprandial hyperglycemia. The investigators expect these studies to show that TRF is effective and sustainable approach to improving metabolic parameters in overweight/obese individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. BMI ≥ 25
3. Stable sleep and work schedule
4. Owns a smart phone
5. Capable of giving informed consent

Exclusion Criteria:

1. Pregnant
2. Nursing
3. Anticipation of pregnancy during the course of the study
4. Clinically significant medical issues as determined by the study clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Weight | 12 weeks
  Change in weight (kg) from baseline to study conclusion

SECONDARY OUTCOMES:
Body composition | 12 weeks
  Change in body composition (% change in body fat as measured by DXA) from baseline to study conclusions

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD, Principal Investigator — University of Minnesota, Division of Diabetes, Endocrinology and Metabolism
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olawsky E, Zhang Y, Eberly LE, Helgeson ES, Chow LS. A New Analysis Tool for Continuous Glucose Monitor Data. J Diabetes Sci Technol. 2022 Nov;16(6):1496-1504. doi: 10.1177/19322968211028909. Epub 2021 Jul 20. PMID 34282646